CLINICAL TRIAL: NCT06137716
Title: Development and Clinical Trials of a Rehabilitation Platform to Accelerate the Recovery of Patients With COVID Neuromotor Sequelae
Brief Title: Robotic Assisted Hand Rehabilitation Outcomes in Adults After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Centro Hospitalario Padre Benito Menni (Unknown)
Responsible Party: Principal Investigator, Juan Carlos Fraile, Professor, University of Valladolid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASVE-NM-22-575
Record Dates: First submitted 2023-11-16; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Robotic Exoskeleton; Post-acute Covid-19 Syndrome; Rehabilitation Outcome; Physical And Rehabilitation Medicine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Experimental): Participants will rehabilitation with a robotic hand exoskeleton.
  Interventions: Device: Training with a Robotic Hand Exoskeleton

INTERVENTIONS:
Device: Training with a Robotic Hand Exoskeleton — The rehabilitation program extended over six consecutive weeks. Each therapy session, lasting 45 minutes, occurred four times per week, resulting in a total of 24 sessions. Within each session, a total of six exercises, consisting of three passive exercises and three bilateral exercises, were performed in an alternating manner. The exercises were executed in the following sequence: 1) Bilateral hand opening and closing; 2) Passive independent finger opening and closing; 3) Bilateral pinch; 4) Passive hand opening and closing; 5) Bilateral hand opening and closing based on a VR-based game involving squeezing an orange; 6) Passive pinch.

SUMMARY:
Prolonged hospitalization in severe COVID-19 cases can lead to substantial muscle loss and functional deterioration. While rehabilitation is vital, conventional approaches encounter capacity constraints. Therefore, assessing the efficacy of robotic-assisted rehabilitation is crucial for post-COVID-19 fatigue syndrome patients, aiming to improve motor function and overall recovery. The study focuses on evaluating rehabilitation effectiveness in individuals with upper-extremity impairment using a hand exoskeleton-based robotic system.

ELIGIBILITY:
Inclusion Criteria:

* Over 30 years old
* Patients infected with COVID-19 and has received care at the Centro Hospitalario Benito Menni
* Patients with acute or limited functional or strength impairment in at least one of the upper extremities
* Patients who would complete a rehabilitation program and a series of patient reported outcome questionnaires and a follow up evaluation
* Patients who give inform written consent.

Exclusion Criteria:

* Presence of behavioral disorders
* Dementia (loss of memory of cognitive functions)
* Disorders of consciousness (confusional states and drowsiness)
* Uncontrolled or severely limiting delusions and hallucinations
* Infectious skin diseases
* Rrisk of epileptic seizures due to COVID itself or prior to it
* Severe visual impairments
* Severe spasticity with a Modified Ashworth Scale >2, joint stiffness in the wrist and fingers
* Pain with a score >8 on the Visual Analog Scale (VAS) during mobilization of the affected hand.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Barthel Index (BI) | Baseline / 6 weeks
  The Barthel Index (BI) modified by Granger et al is an ordinal scale for measuring the ability of an individual to independently execute 15 activities of daily living (ADL) related with mobility and self-care. BI aims to evaluate the degree of independence, with a final score ranging from 0 to 100, where 0 indicates full dependence.
Functional Independence Measure (MIF) | Baseline / 6 weeks
  The Functional Independence Measure (MIF) was designed to provide an indicator of disability independent of a patient's impairment. The scale consists of 18 items to evaluate functional abilities in the area of communication, locomotion, self-care, social cognition, sphincter control and transfers. Each of these items is quantified utilizing a 7-point Likert scale. The total score, obtained by summing the individual item scores, spans from 18 to 126, with 18 denoting a state of complete dependence
SF-36 Health Questionnaire | Baseline / 6 weeks
  The SF-36 Health Questionnaire consists of 36 items designed to assess health-related quality of live. It encompasses eight scales, each comprising 2 to 10 items, which aimed to evaluate various health attributes. These scales include physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health.The score of each scale ranges from 0 to 100, with higher scores indicating a better health-related quality of life.
Range of motion | Baseline / 6 weeks
  The range of motion was analyzed by goniometry measurements using the HandTutor® glove. It provides the active and passive movement of the participants fingers through sensors located in the front and back of the glove.

SECONDARY OUTCOMES:
Semi-structured interview | Baseline
  Additional information about personal and environmental factors and participatio

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalario Padre Benito Menni, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cisnal A, Alonso-Linaje G, Fraile JC, Perez-Turiel J, Alvarez P, Martinez S. Tackling Post-COVID-19 Rehabilitation Challenges: A Pilot Clinical Trial Investigating the Role of Robotic-Assisted Hand Rehabilitation. J Clin Med. 2024 Mar 7;13(6):1543. doi: 10.3390/jcm13061543. PMID 38541769